CLINICAL TRIAL: NCT05020821
Title: Superior Trunk Block Catheter Versus Single-shot Superior Trunk Block With Intravenous Dexmedetomidine for Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2021-0853
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Arthroplasty; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-shot superior trunk block with intravenous dexmedetomidine (Active Comparator): participants receiving single-shot superior trunk block with intravenous dexmedetomidine
  Interventions: Procedure: Single-shot superior trunk block with intravenous dexmedetomidine
- Continuous superior trunk block (Experimental): participants receiving continuous superior trunk block
  Interventions: Procedure: Continuous superior trunk block

INTERVENTIONS:
Procedure: Single-shot superior trunk block with intravenous dexmedetomidine — During surgery, dexmedetomidine will be administered. After intravenous administration of 2 mcg/kg for 30 minutes, 0.5 mcg/kg/hr will be administered until the end of surgery. After surgery, a single-shot superior trunk block will be performed under ultrasound guidance. 15 mL of 0.5% ropivacaine with 1:200,000 epinephrine will be administered.
  Arms: Single-shot superior trunk block with intravenous dexmedetomidine
Procedure: Continuous superior trunk block — During surgery, an equivalent volume of the placebo solution was administered in a similar manner as dexmedetomidine. The superior trunk block catheter will be inserted under ultrasound guidance using 15 mL of 0.5% ropivacaine after the operation and utilize patient-controlled analgesia infusion pump with a 300 mL reservoir of ropivacaine 0.2%, and programmed the pump to deliver 5 mL per hour with an optional patient-controlled analgesia bolus of 4 mL at 30-minute lockout intervals. Patients were typically discharged home on POD 1, and block was continued until reservoir completion.
  Arms: Continuous superior trunk block

SUMMARY:
Shoulder arthroplasty is associated with significant postoperative pain. Appropriate pain control after shoulder arthroplasty is crucial for postoperative rehabilitation and patient satisfaction. Superior trunk block is a commonly employed regional anesthetic technique for shouler arthroplasty, and a continuous catheter is often placed to extend the analgesic benefit of the block. However, continuous peripheral nervel block (PNB) is more costly and time-consuming than sigle-shot PNB. Recent evidence suggests that intravenous (IV) dexmedetomidine (DEX) prolong the analgesic duration after sigle-shot PNB. The investigators will compare continuous superior trunk block with single-shot superior trunk block with IV DEX in patients undergoing shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1 Patients aged 19 years old or older, with American Society of Anesthesiologists Physical Status 1-3, and scheduled for elective shoulder arthroplasty

Exclusion Criteria:

1. Allergy or intolerance to any of the drugs used in the study
2. Heart failure
3. Hepatic or renal insufficiency
4. Opioid dependency
5. Coagulopathy
6. Pre-existing neurologic or anatomic deficits in the upper extremities
7. Severe psychiatric illness

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale pain score | 24 hours after the end of surgery
  Pain intensity at rest will be evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) 24 hours after the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No